CLINICAL TRIAL: NCT06393842
Title: Correlation of the Non-invasive Cardiopulmonary Management Wearable Device With Measures of Congestion in Heart Failure in Exercise - CONGEST - HF - EX
Brief Title: Correlation of Non-invasive CPM Wearable Device With Measures of Congestion in Heart Failure in Exercise
Acronym: CONGEST-HFEX
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Analog Devices (Unknown)
Responsible Party: Sponsor
Other Study IDs: INGN22CA411
Record Dates: First submitted 2024-02-19; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Pulmonary Congestion
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cohort A: Patients receiving hemodialysis: Primary Objective is to investigate if changes in measures derived by the CPM wearable device correlate with changes in B-lines between dialysis sessions and with the difference in weight between dialysis sessions. The end point would be to demonstrate a change in number of B-Lines on Lung Ultrasound between dialysis sessions and compare it with changes in measures derived by CPM wearable device (thoracic impedance and S3) taken during the same sessions. We would then use correlation coefficient to find how strong a relationship is between measures from Lung Ultrasound and CPM wearable device.
  Secondary objective will include correlation of the measures from CPM wearable device with other measures of congestion including Spirometry, Echocardiography, Biomarkers and Physical symptoms and signs including EVEREST and ASCEND congestion score
  Interventions: Device: Cardiopulmonary Management Wearable Device
- Cohort B: Primary Objective- Patients receiving inpatient intravenous diuretic treatment for heart failure. To investigate if measures derived by the CPM wearable device system correlate with B-lines on lung ultrasound before and after exercise during the treatment for HF. The end point would be to demonstrate a change in number of B-Lines on LUS before and after exercise during decongestion treatment for HF and compare it with measures derived by CPM wearable device (thoracic impedance and S3) taken during the same sessions. We would then use correlation coefficient to find how strong a relationship is between measures from LUS and CPM wearable device and whether the correlation improved following exercise.
  Secondary objective will include correlation of the measures from CPM wearable device with other measures of congestion including Spirometry, Echocardiography, Biomarkers and Physical symptoms and signs including EVEREST and ASCEND congestion score
  Interventions: Device: Cardiopulmonary Management Wearable Device

INTERVENTIONS:
Device: Cardiopulmonary Management Wearable Device — Fluid status and congestion can be determined by the CPM wearable device and correlates with non-invasive measures and biochemical markers of congestion and changes in congestion.

SUMMARY:
Fluid status and congestion can be determined by the CPM wearable device and correlates with non-invasive measures and biochemical markers of congestion and changes in congestion.

DETAILED DESCRIPTION:
Heart Failure is common, affecting 1-2% of the general population, with the prevalence increasing to over 10% in those over the age of 80. Heart Failure is associated with high morbidity, with many patients requiring frequent and often lengthy hospitalization for treatment with intra venous diuretics. In the recent Heart Failure audit of England and Wales, of over 68000 patients admitted to hospital with a primary diagnosis of Heart Failure between 2017 and 2018, median length of stay was 6-9 days, depending on whether patients were managed by specialist cardiologists. Heart Failure hospitalizations account for approximately 5% of all emergency admissions leading to 2% of all NHS inpatient bed-days. Heart Failure accounts for almost 2% of the total NHS budget, with approximately 70% of these costs due to Heart Failure hospitalizations. The hallmark of decompensation is the development of congestion. This is usually manifested by the development or worsening of pulmonary edema or peripheral edema. Patients often present to hospital when the degree of congestion becomes severe enough to cause symptoms, most often shortness of breath, and therefore require treatment through decongestion with vasodilators and intra venous diuretics. However, a number of studies have shown that the presence of congestion can be detected days to weeks prior to hospitalization leaving a window of opportunity in which treatment aimed at averting a costly hospitalization could occur. Furthermore, congestion can be altered by exercise and may be more pronounced on exercise. Detecting these early signs of congestion has so far only been possible using invasive monitoring devices such as specially designed pacemakers (Heart Logic™, Boston Scientific) or implantable pressure monitors (Cardio MEMS™, Abbott)

Analog Devices Inc have developed a wearable patch-like device called the Cardio- Pulmonary Management (CPM) wearable device which is applied to a patient's chest to assess congestion levels by measuring a number of physiological parameters over approximately five minutes. The goal of this Prospective Uncontrolled Clinical Investigation is to determine if the CPM wearable device can accurately detect the presence of congestion by correlating the findings from the device with changes in congestion status in patients receiving hemodialysis (Cohort A) and if the correlations are different before and after exercise in patients receiving treatment for decongestion for heart failure as an inpatient (Cohort B) as measured by lung spirometry, lung ultrasound Trans Thoracic Echocardiography and Biomarkers

ELIGIBILITY:
Inclusion Criteria:

Written informed consent Male or female ≥18 years of age

Cohort A

1. Established on hemodialysis for >90 days
2. Undergoing hemodialysis with target volume removal ≥1.5 liters fluid

Cohort B Meet ESC criteria for diagnosis of Heart Failure including

1. Heart failure with reduced (HF-REF), mid-range (HF-mREF) and preserved (HF-PEF) ejection fractions
2. Requiring treatment with intravenous (IV) diuretics

Exclusion Criteria:

1. Unable to consent to inclusion in study due to cognitive impairment
2. Allergies or skin sensitivities to silicone- based adhesive
3. Skin breakdown or dermatological condition on the left chest or breast areas or chest wall deformity where the device is placed
4. Pregnancy or breast-feeding
5. Currently uncontrolled cardiac arrhythmia
6. Hemodynamically significant mitral stenosis (at least moderate in severity on TTE)
7. Conditions that may confound congestion assessments including

A. Severe obstructive lung disease B. Severe fibrotic lung disease C. Severe liver disease D. Relevant active malignancy E. Active viral or bacterial bronchopneumonia-CXR within 4 weeks showing consolidation F. Pulmonary contusion G. Pneumothorax H. Pneumonectomy I. Lobectomy J. Pulmonary embolism within the previous 3 months K. Indwelling intercostal chest drain L. Left ventricular assist device (LVAD) M. COVID-19 infection. N. Increased Body Mass Index where satisfactory Echocardiographic images not possible

Cohort B only - inability to perform exercise safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A- Dialysis patients (Inpatients and Outpatients) at the Queen Elizabeth University Hospital, Glasgow
  Cohort B- Heart Failure Hospitalizations at the Queen Elizabeth University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-02-06 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
To investigate if changes in measures derived by the CPM wearable device correlate with changes in B-lines between dialysis sessions and with the difference in weight between dialysis sessions. | Between Two Consecutive Dialysis Session (Day 1 and Day 3)
  Correlation of change in congestion measured by the CPM wearable device (thoracic impedance and S3) and change in lung ultrasound (LUS) and weight between the end of the dialysis session and the start of the subsequent dialysis session in patients undergoing two consecutive hemodialysis sessions.
To investigate if measures derived by the CPM wearable device system correlate with B-lines on lung ultrasound before and after exercise during the treatment for HF. | Data will be gathered at four time points: (1) on the day of enrolment; (2) the day after enrolment; (3) within 24 hours of switch from IV to oral diuretics and; (4) when the patient is as euvolemic as reasonably achievable
  To compare correlations of congestion measured by the CPM wearable device (thoracic impedance and S3) and clinical measures of congestion (LUS) in inpatients with HF obtained before and after exercise

SECONDARY OUTCOMES:
To determine the correlation between change in pulmonary function measured by the CPM wearable device and change in pulmonary function measured with spirometry between two consecutive dialysis sessions. | Between Two Consecutive Dialysis Session (Day 1 and Day 3)
  To determine the correlation between change in pulmonary function measured by the CPM device (tidal volume) and pulmonary function measured with spirometry between the end of the dialysis session and the start of the subsequent dialysis session in patients undergoing two consecutive hemodialysis sessions.
  To determine the correlation between change in congestion measured by the CPM wearable device (thoracic impedance and S3) and change in clinical measures of congestion [physical symptoms and signs and TTE findings] between the end of the dialysis session and the start of the subsequent dialysis session in patients undergoing two consecutive hemodialysis sessions.
To compare the correlations, before and after exercise, between congestion measured by the CPM wearable device (thoracic impedance and S3) and TTE findings. | Data will be gathered at four time points: (1) on the day of enrolment; (2) the day after enrolment; (3) within 24 hours of switch from IV to oral diuretics and; (4) when the patient is as euvolemic as reasonably achievable
  The end point would be to demonstrate change in IVC size and change in parameters such as TR Vmax and E/e' on Echocardiography before and after exercise during decongestion treatment for HF and compare it with change in congestion measured by CPM wearable device during the same sessions. We would then use correlation coefficient to find how strong a relationship is between echocardiographic parameters and CPM wearable device.

CONTACTS AND LOCATIONS:
Overall Officials: Pardeep Jhund, FRCP, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Glasgow Cardiovascular Research Centre, Glasgow, Scotland, United Kingdom